CLINICAL TRIAL: NCT07001995
Title: A Single-center, Single-arm Phase II Study of Limertinib Plus Carboplatin and Etoposide in EGFR-mutant NSCLC Patients With SCLC Transformation After EGFR-TKI Progression
Brief Title: Limertinib Plus Carboplatin and Etoposide for EGFR-mutant NSCLC With SCLC Transformation After EGFR-TKI Progression
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Director, Head of Medical Oncology, Principal Investigator, Clinical Professor, Hunan Province Tumor Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALLISTO
Record Dates: First submitted 2025-05-25; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Small Cell Lung Cancer; Non Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Etoposide; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Limertinib Carboplatin Etoposide
  Interventions: Drug: limertinib; Drug: etoposide and carboplatin

INTERVENTIONS:
Drug: limertinib — limertinib 80 mg
Drug: etoposide and carboplatin — etoposide 100 mg/m² IV D1-3 + carboplatin AUC 5-6 IV
  Other Names: EC

SUMMARY:
This single-center, prospective study and aims to evaluate the efficacy and safety of limertinib combined with etoposide and carboplatin in EGFR-mutant NSCLC patients who develop small-cell lung cancer transformation following progression on EGFR-TKI therapy.

DETAILED DESCRIPTION:
This is a single-center, prospective interventional Phase II study designed to assess the efficacy, safety and mechanism of resistance to limertinib combined with carboplatin and etoposide in EGFR-mutant NSCLC patients who have histologically confirmed small-cell transformation after progression on EGFR-TKI therapy. Thirty patients will receive Limertinib orally once daily (80 mg) plus carboplatin (AUC 5-6, day 1) and etoposide (100 mg/m², days 1-3) every 21 days until disease progression or unacceptable toxicity. Radiographic tumor evaluation will be conducted every 6 weeks per RECIST v1.1. Tumor tissue and blood specimens will be collected at baseline and upon disease progression for next-generation sequencing to elucidate the molecular mechanisms underlying histological transformation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following to be eligible for enrollment:
* Signed written informed consent prior to any study-related procedures.
* Age ≥ 18 and ≤ 80 years.
* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) with a sensitizing EGFR mutation (exon 19 deletion or L858R, with or without concurrent mutations).
* Prior treatment with EGFR-TKI, with documented disease progression and histologically confirmed small-cell lung cancer (SCLC) transformation.
* At least one measurable target lesion per RECIST v1.1.
* ECOG performance status 0-1 (see Appendix for ECOG scale).
* Estimated life expectancy > 3 months.
* Adequate bone marrow function, defined as:
* ANC ≥ 1,500/mm³
* Hemoglobin ≥ 9 g/dL
* Platelets ≥ 90,000/mm³
* Adequate hepatic function, defined as:
* Total bilirubin ≤ 1.5 × ULN
* AST and ALT ≤ 2.5 × ULN (or ≤ 5 × ULN in patients with known hepatic metastases)
* Adequate renal function, defined as:
* Serum creatinine within normal limits OR creatinine clearance ≥ 50 mL/min (Cockcroft-Gault)
* For patients with BMI < 18.5 or > 30, eGFR ≥ 50 mL/min (MDRD) is acceptable
* Adequate cardiac function, defined as LVEF ≥ 50% by MUGA scan or echocardiography.
* Women of childbearing potential and men with partners of childbearing potential must agree to use effective contraception.

Exclusion Criteria:

* Patients meeting any of the following criteria will be excluded from the study:
* Histology at initial diagnosis of small-cell lung cancer (SCLC), large-cell carcinoma, or mixed tumor with predominant SCLC, large-cell, or neuroendocrine components.
* Prior treatment with a standard SCLC chemotherapy regimen (e.g., carboplatin/etoposide or cisplatin/etoposide) after SCLC transformation.
* Symptomatic or unstable brain metastases. Patients with a history of unstable brain metastases must have undergone definitive surgery or radiotherapy, remain clinically stable, and be off corticosteroids for cerebral edema for at least 14 days before enrollment.
* Any concurrent malignancy other than basal cell carcinoma of the skin or carcinoma in situ of the cervix. (Patients with a prior malignancy must be disease-free for ≥ 5 years to be eligible.)
* Pregnancy (confirmed by serum ß-hCG) or breastfeeding. Note: Women who have been postmenopausal for ≥ 12 months, or who have undergone hysterectomy, bilateral oophorectomy, or bilateral tubal ligation, are exempt from contraception requirements. Male participants must use effective contraception from the first dose of study drug until 180 days after the last dose.
* Active hepatitis B (HBV DNA > 1,000 IU/mL) or hepatitis C infection (anti-HCV positive and/or HCV RNA > 15 IU/L), or known HIV infection.
* Known hypersensitivity to lietinib, carboplatin, or etoposide.
* Psychiatric or cognitive disorders that would preclude informed consent or compliance with study requirements.
* Women planning pregnancy during the screening period or who, along with their partners, are not using effective contraception.
* Any other medical or psychosocial condition judged by the investigator to compromise patient safety or study integrity (e.g., poor compliance or comorbidities affecting efficacy assessment).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Time from first subject dose to study completion, or up to 36 month
  define as first dose to first documented disease progression assessed by investigator or death due to any cause

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Time from first subject dose to study completion, or up to 36 month
  According to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator, define as the proportion of subjects who have a complete response (CR) or a partial response (PR)
Disease control response (DcR) | Time from first subject dose to study completion, or up to 36 month
  According to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator, define as the proportion of subjects who have a complete response (CR) , partial response (PR) or stable disease (SD)
Duration of Response (DoR) | Time from first subject dose to study completion, or up to 36 month
  To assess duration of response for subjects with CR or PR according to RECIST version 1.1 by investigator , defined as the time from the first documented CR or PR to disease progression or death
Adverse events (AEs) | From first dose to the last dose, up to 24 month
  Number of participants with adverse events (AEs) according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Yongchang Zhang, Changsha, Hunan, China